CLINICAL TRIAL: NCT03469297
Title: Early Feasibility Study of the Brown Glaucoma Implant in Patients With No Light Perceived
Brief Title: Early Feasibility Study of the Brown Glaucoma Implant in Patients With Severe Visual Impairment or No Light Perceived
Acronym: Early Bird
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroOptx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4039
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Results first posted 2022-12-05 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Brown Glaucoma Implant (Experimental)
  Interventions: Device: Brown Glaucoma Implant

INTERVENTIONS:
Device: Brown Glaucoma Implant — The Brown Glaucoma Implant (BGI) is an implantable device designed to lower intraocular pressure (IOP) in glaucoma patients by shunting aqueous humor from the anterior chamber of the eye to the surface of the eye. Because there are no physiologic sources of outflow resistance, the device can be engineered to target an IOP that is low enough to halt the progression to blindness in a patient suffering from glaucoma.

SUMMARY:
This is a prospective, non-randomized, single-arm early feasibility study to assess the safety and feasibility of lowering intraocular pressure with the Brown Glaucoma Implant. A total of up to 10 subjects will be enrolled at three centers. Subjects will be followed for 24 months, with the primary assessments completed 6 months after implant.

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 years and older.
2. Best corrected visual acuity of 20/400 or worse.in the study eye.
3. Fellow eye with visually acuity of 20/200 or better and the visual field no worse than the study eye. If the study eye has no light perception, the fellow eye may have no light perception or better.
4. Intraocular pressure in the study eye greater than or equal to 21 mmHg and less than or equal to 50 mmHg.
5. Primary open-angle glaucoma (confirmed by gonioscopy).
6. Glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities: (1) Diffuse thinning, focal narrowing, or notching of the optic disc rim, especially at the inferior or superior poles with or without disc hemorrhage; (2) Localized abnormalities of the peripapillary retinal nerve fiber layer, especially at the inferior or superior poles; or (3) Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue.
7. Humphrey Visual Field (HVF) demonstrating visual field defects consistent with glaucomatous optic nerve damage.
8. At least two contiguous clock hours of intact conjunctiva near the limbus between clock hours of 9:00 and 03:00 in the study eye.
9. Adequate space in the anterior chamber of the study eye sufficient to support implant with the BGI, defined as two contiguous clock hours of scleral spur visualization via goinioscopy, without compression, in the superior 180 degrees of the anterior angle.
10. Able and willing to comply with protocol requirements.
11. Able to understand and sign the Informed Consent form.

Exclusion Criteria:

1. Active Neovascular Glaucoma in the study eye.
2. Pigmentary Glaucoma in the study eye.
3. Pseudoexfoliative Glaucoma in the study eye.
4. Corneal conditions in the study eye that may inhibit normal incisional healing (e.g. Fuch's dystrophy) or impair visualization of the implant inside the anterior chamber.
5. Anticipated need for ocular surgery within one year in the study eye.
6. Requirement of a combined glaucoma procedure in the study eye.
7. Contact lens use in the study eye.
8. Clinically significant inflammation or infection in the study eye within 60 days prior to the preoperative visit (e.g., blepharitis, conjunctivitis, keratitis, uveitis, herpes simplex infection) or any systemic infection. For purposes of this study, clinically significant is considered any such condition requiring prescription therapy.
9. Other clinical conditions:

   1. Poorly controlled diabetes (Type I or Type II) as determined by HbA1c >8.
   2. Cancer requiring treatment during the duration of the study.
   3. Any drugs (e.g.: immunosuppressive drugs) or co-morbidity that might inhibit wound healing.
10. Participation in any other clinical trial during participation in this trial.
11. Life expectancy <1 year.

If both eyes of a prospective trial participant are eligible, only the eye with the highest intraocular pressure will be selected for implant.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2021-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Minnesota Eye Consultants, Bloomington, Minnesota
  - iWorks Laser and Vision Center, Dayton, Ohio
  - Glaucoma Associates of Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brown Glaucoma Implant
Started | 8 (Implanted)
Completed | 7 (Completed 6 months of follow-up)
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: 8 subjects were consented and implanted. 7 subjects completed the Month 6 post-implant visit and were included in endpoint analyses. 5 subjects completed the study with 24 months of follow-up post-implant.
Arm/Group | Brown Glaucoma Implant
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Responder Rate
Description: Responder rate defined as achieving at least 20% reduction from baseline in intra-ocular pressure (IOP)
Time Frame: 6 Months
Population: Implanted subjects completing the 6-month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Brown Glaucoma Implant
Number analyzed (Participants) | 7
Participants | 3

2. Primary Outcome: Adverse Event Rate
Description: Rate of all AEs
Time Frame: 6 Months
Population: Implanted subjects
Measure: Number; unit: Events
Arm/Group | Brown Glaucoma Implant
Number analyzed (Participants) | 7
Events
  Adverse Events | 66
  Serious Adverse Events | 8
  Device-Related Adverse Events | 31
  Procedure-Related Adverse Events | 12

3. Secondary Outcome: Mean Change From Baseline in IOP
Description: Mean change in diurnal IOP since the baseline visit
Time Frame: Baseline, 6 Months
Population: Implanted subjects completing the 6-month visit.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Brown Glaucoma Implant
Number analyzed (Participants) | 7
mmHg | 8.3 (14.9)

4. Secondary Outcome: Alternative Responder Rate
Description: Responder rate defined as achieving follow-up IOP less than or equal to 14mmHg
Time Frame: 6 Months
Population: Implanted subjects who completed the month 6 follow-up visit
Measure: Count of Participants; unit: Participants
Arm/Group | Brown Glaucoma Implant
Number analyzed (Participants) | 7
Participants | 3

5. Secondary Outcome: Change in IOP-lowering Medications
Description: Mean change in number of glaucoma medications since baseline
Time Frame: Baseline, 6 Months
Population: Implanted subjects who completed the month 6 follow-up visit
Measure: Mean (Standard Deviation); unit: Number of Glaucoma Medications
Arm/Group | Brown Glaucoma Implant
Number analyzed (Participants) | 7
Number of Glaucoma Medications | 0.6 (1.8)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Brown Glaucoma Implant
All-Cause Mortality (participants affected / at risk) | 2/7
Serious Adverse Events (participants affected / at risk) | 4/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brown Glaucoma Implant (N=7)
Atypical Chest Pain (Cardiac disorders) | 1 (1)
Mental Health Crisis Evaluation (Psychiatric disorders) | 1 (1)
Increased Intra-Ocular Pressure (Eye disorders) | 1 (1) — In non-study eye
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left Knee Replacement (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brown Glaucoma Implant (N=7)
Anterior Chamber Flare (Eye disorders) | 1 (2)
Blurred Vision (Eye disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Chalazion (Eye disorders) | 1 (1)
Choroidal Detachment (Eye disorders) | 1 (1)
Conjunctivitis/Conjunctival Injection (Eye disorders) | 5 (8)
Corneal Abrasion (Eye disorders) | 2 (2)
Corneal Edema (Eye disorders) | 1 (1)
Diminished/No Flow through BAM Device Channel (Eye disorders) | 3 (9)
Eye Dryness/Discomfort/Irritation (Eye disorders) | 2 (5)
Epistaxis (General disorders) | 1 (1)
Folliculitis - Trunk (Skin and subcutaneous tissue disorders) | 1 (1)
Increased Intra-Ocular Pressure (Eye disorders) | 6 (12)
Iris Nevus (Eye disorders) | 1 (1)
Knee Surgery (Surgical and medical procedures) | 1 (1)
Migraine Headache (General disorders) | 1 (1)
Ocular Allergies (Eye disorders) | 2 (3)
Posterior Capsular Opacification (Eye disorders) | 1 (1)
Bleeding During Implant Procedure (Surgical and medical procedures) | 1 (1)
Sinusitis (General disorders) | 1 (3)
Skin Lesion - Forearm (Injury, poisoning and procedural complications) | 1 (1)
Superficial Punctate Keratitis (Eye disorders) | 2 (3)
Tenon Cyst (Eye disorders) | 1 (1)
Unilateral Icteric Sclera (Eye disorders) | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vessels on Endothelium (Eye disorders) | 1 (1)
Eye Watering (Eye disorders) | 1 (1)
Eye Feels Tired (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Approximately 2 weeks after the initial implant, one subject (02-03) had the first BAM device explanted due to device channel blockage and elevated intra-ocular pressure. A second BAM device was implanted immediately after the explant procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-01-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT03469297/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT03469297/SAP_001.pdf